CLINICAL TRIAL: NCT04481009
Title: A Multicenter, Open-Label, Phase I/II Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of YH003 in Combination With Toripalimab (Anti-PD-1 mAb) in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate YH003 in Combination With Toripalimab (Anti-PD-1 mAb) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YH003002
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — toripalimab; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YH003 with Toripalimab after PD-1/L1 +/- CTLA-4 treatment (Experimental): YH003 in combination with Toripalimab in subjects with unresectable /metastatic melanoma after having failed PD-1/L1 +/- CTLA-4 treatment.
  Interventions: Drug: YH003; Drug: Toripalimab
- YH003 with Toripalimab in subjects with PDAC (Experimental): YH003 in combination with Toripalimab in subjects with unresectable/ metastatic pancreatic ductal adenocarcinoma (PDAC) as 2nd line treatment.
  Interventions: Drug: YH003; Drug: Toripalimab
- YH003 with Toripalimab plus standard chemotherapy (Experimental): YH003 in combination with Toripalimab plus standard chemotherapy (Nab-paclitaxel + Gemcitabine) in subjects with unresectable/metastatic PDAC as 1st line treatment
  Interventions: Drug: YH003; Drug: Toripalimab; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: YH003 — YH003 will be administered intravenously over 60 minutes every 21-day cycle.
Drug: Toripalimab — Toripalimab with fixed dose of 240 mg administered intravenously followed by YH003 administered intravenously every 21-day cycle.
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered each 21-day cycle.
  Arms: YH003 with Toripalimab plus standard chemotherapy
Drug: Gemcitabine — Gemcitabine will be administrated each 21-day cycle.
  Arms: YH003 with Toripalimab plus standard chemotherapy

SUMMARY:
This is a phase I/II, multi-center, open-label study of YH003 in combination with Toripalimab (anti-PD-1 mAb). The study is comprised of a dose escalation part (Part I) exploring escalating doses of YH003 in combination with fixed dose toripalimab in subjects with advanced solid tumors (Part I), followed by an expansion part (Part II) with three expansion cohorts.

DETAILED DESCRIPTION:
The study is comprised of a dose escalation part (Part I) exploring escalating doses of YH003 in combination with fixed dose toripalimab in subjects with advanced solid tumors (Part I), followed by an expansion part (Part II) with three expansion cohorts.

During Part I, dose escalation part of the study, a traditional 3+3 dose algorithm will be utilized to identify MTD(maximum tolerated dose) and/or RP2D (recommended phase 2 dose).

This dose escalation part will consist two phases, the run-in phase to explore safety and tolerability of YH003 as single agent and the combination phase to explore safety and tolerability of escalating doses of YH003 in combination with fixed dose Toripalimab.

The Phase II expansion part of this clinical trial will include three parallel cohorts(cohort 2A, 2B and 2C) of 20 subjects each treated with a dose around the RP2D of YH003 in combination with Toripalimab to assess the antitumor activity and safety/tolerability. One expansion cohort (2A) is YH003 and toripalimab in subjects with unresectable/metastatic melanoma, the other two expansion cohorts (2B and 2C) are YH003 and toripalimab with or without nab-paclitaxel + gemcitabine in unresectable/ metastatic pancreatic ductal adenocarcinoma.

Subjects will be monitored for safety, tolerability and efficacy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the ability to understand and willingness to sign a written informed consent document.
2. Part I dose escalation:

   Have histologically advanced or cytologically confirmed solid tumor. Have progressed on after treatment with at least one standard therapy or intolerant of the standard therapy.

   Part II dose expansion:

   Cohort 2A: Histologically or cytologically confirmed unresectable or metastatic melanoma that had confirmed progressive disease during treatment with an anti-PD-1/PD-L1 therapy with or without additional CTLA-4 therapy. Subjects with BRAF activating mutation could have also received a BRAF inhibitor and/or MEK inhibitor regimen prior to anti-PD-1/PD-L1 therapy.

   Cohort 2B, 2C: Subject has histologically or cytologically documented diagnosis of pancreatic ductal adenocarcinoma with unresectable locally advanced/metastatic disease Cohort 2B: had confirmed progressive disease during treatment with first line standard of care of chemotherapy per local standard.

   Cohort 2C: treatment-naïve for unresectable locally advanced/metastatic disease.
3. Subject must have measurable disease by RECIST 1.1. At least 1 unidimensional measurable target lesion per RECIST v1.1 for study Part II expansion cohorts.
4. Subjects must be age 18 years or older.
5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Life expectancy ≥3 months.
6. Subjects must have adequate organ function.
7. Women of reproductive potential must have negative serum beta human chorionic gonadotropin (β -HCG) pregnancy test.

Exclusion Criteria:

1. Part II Cohort 2A: History of life-threatening toxicity or treatment discontinuation due to related to prior anti-PD-1/PD-L1 and with or without CTLA-4 combination treatment for subjects with unresectable/metastatic melanoma.
2. Subjects must not have another active invasive malignancy.
3. Previous exposure to TNFR such as anti-CD137, OX40, CD27 and CD357 antibodies.
4. Subjects must not have received any anticancer therapy or another investigational agent within the shorter of 4 weeks or 5 half-lives before the first dose of the study treatment.
5. Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy.
6. History of clinically significant sensitivity or allergy to monoclonal antibodies and their excipients or known allergies to antibodies produced from Chinese hamster ovary cells, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to YH003 or Toripalimab. Also history of severe hypersensitivity reaction to Nap-paclitaxel and/or gemcitabine.
7. Primary central nervous system (CNS) malignancies or symptomatic CNS metastases.
8. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease.
9. Subjects must not have a known or suspected history of an autoimmune disorder, including but not limited to inflammatory bowel disease, celiac disease, Wegner syndrome, Hashimoto syndrome, systemic lupus erythematosus, scleroderma, sarcoidosis, or autoimmune hepatitis, within 3 years of the first dose of study treatment.
10. Clinically uncontrolled intercurrent illness, including an ongoing or active infection, active coagulopathy, uncontrolled diabetes, psychiatric illness that would limit compliance with the study requirements and other serious medical illnesses requiring systemic therapies.
11. Severe cardiovascular disease including symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina, uncontrolled hypertension, cardiac arrhythmia, a history of myocardial infarction within 6 months or a history of arterial thromboembolic event and pulmonary embolism within 3 months of the first dose of investigational agent.
12. QTc > 450 ms at baseline; no concomitant medications that would prolong the QT interval; no family history of long QT syndrome.
13. Subjects must not have active infection of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
14. Subjects must not have a history of primary immunodeficiency.
15. Subjects from endemic area will be specifically screened for tuberculosis. Subjects with active tuberculosis are excluded.
16. Subjects must not receive concurrent or prior use of an immunosuppressive agent within 4 weeks of the first dose of YH003.
17. Major surgery within 4 weeks prior to study entry and Minor surgery within 2 weeks prior to the first dose of YH003.
18. Subjects must not have received a live attenuated vaccine within 28 days before the first dose of YH003, and subjects, if enrolled, should not receive live vaccines during the study or for 180 days after the last dose of YH003.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Overall safety and tolerability profile of YH003 in combination with Toripalimab. | From screening up to 1 year
  The safety profile of YH003 in combination with Toripalimab will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0
Maximum tolerated dose (MTD) and Recommended phase 2 dose (RP2D) | Cycle 1 of each cohort. Duration of one cycle is 3 weeks
  The MTD and RP2D will be determined based on the data of safety and tolerability

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Maximum serum concentration (Cmax) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Trough concentration before the next dose is administered (Ctrough) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Time to reach maximum serum concentration (Tmax) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Clearance (CL) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Volume of distribution (Vd) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Volume of distribution at steady state (Vss) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Terminal half-life (T1/2) | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Dose proportionality | Up to 1 year
  To determine the PK profile of YH003 alone and in combination with Toripalimab
Incidence of anti-drug antibodies (ADAs) | Up to 1 year
  To assess the immunogenicity of YH003 in combination with Toripalimab
Incidence of neutralizing antibodies (NAbs) | Up to 1 year
  To assess the immunogenicity of YH003 in combination with Toripalimab
Objective response rate (ORR) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab
Duration of response (DOR) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab
Time to response (TTR) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab
Progression free survival (PFS) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab
Overall survival (OS) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab
Disease control rate (DCR) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab
Duration of disease control (DDC) | Up to 1 year
  To assess the preliminary antitumor activity of YH003 in combination with Toripalimab

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia